CLINICAL TRIAL: NCT04196296
Title: Brief Online Interventions to Facilitate Treatment Seeking for Social Anxiety
Brief Title: Treatment Seeking for Social Anxiety
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Boulder (Other)
Responsible Party: Principal Investigator, Joanna Arch, Associate Professor, Department of Psychology and Neuroscience, University of Colorado, Boulder
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 15-0452
Record Dates: First submitted 2019-11-27; First posted 2019-12-12 (Actual); Last update posted 2019-12-12 (Actual); Status verified 2019-12

CONDITIONS: Social Anxiety
MeSH Terms: interventions — Information Motivation Behavioral Skills Model

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Psychoeducation (Active Comparator)
  Interventions: Behavioral: Psychoeducation
- Psychoeducation plus Motivation Enhancement (Experimental)
  Interventions: Behavioral: Psychoeducation; Behavioral: Motivation

INTERVENTIONS:
Behavioral: Psychoeducation — Online psychoeducation about social anxiety, evidence-based treatments that target social anxiety, and treatment referral/resource information.
Behavioral: Motivation — Online exercises/activities regarding social anxiety (and treatment thereof) based in principles from Acceptance and Commitment Therapy (ACT) and Motivational Interviewing (MI)/Motivational Enhancement Therapy (MET).
  Arms: Psychoeducation plus Motivation Enhancement

SUMMARY:
This study developed and then compared via randomized trial two brief online interventions targeting increasing treatment-seeking behavior in social anxiety.

ELIGIBILITY:
Inclusion Criteria:

* High social anxiety (score >30 on Social Phobia Inventory (SPIN) Connor et al., 2000)
* Fluent in English
* Amazon Mechanical Turk HIT approval rate > 95%
* Amazon Mechanical Turk account listed as US resident

Exclusion Criteria:

* Already enrolled in target treatments (i.e. CBT for social anxiety, using social anxiety self-help book, or participating in online treatment for social anxiety)
* Indicating that they would "never consider" treatment for social anxiety

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 919 (Actual)
Dates: Start 2016-03-28 (Actual); Primary Completion 2016-07-06 (Actual); Study Completion 2016-07-06 (Actual)

PRIMARY OUTCOMES:
Treatment seeking motivations: Attitudes toward seeking treatment for social anxiety. | Change from baseline to one-month follow-up
  Affective attitudes toward seeking treatment for social anxiety were assessed using a standard 7-item 1-7 semantic differential scale in which participants rated "seeking treatment for social anxiety in the next month would be" according to opposite adjective pairs (e.g., "Unhealthy"/"Healthy"). Possible scores range from 7-49, with higher scores indicating more favorable attitudes toward seeking treatment for social anxiety.
Treatment seeking motivations: Intentions to seek treatment for social anxiety. | Change from baseline to one-month follow-up
  As the existing literature lacks a sufficient and specific scale for assessing intentions to seek treatment, we developed a scale based on the Theory of Planned Behavior (https://doi.org/10.1016/0749-5978(91)90020-T) as well as crucial steps toward seeking treatment identified previously (https://doi.org/10.1016/S0887-6185(02)00259-1). The resulting scale includes 13 total items assessing intentions to seek treatment for social anxiety in the following month. Items were rated using Likert scales from 1 ("strongly disagree"/"not very likely") to 7 ("strongly agree"/"very likely"), with higher scores indicating greater intention to seek treatment for social anxiety within the following month.
Treatment seeking motivations: Perceived behavioral control/confidence regarding seeking treatment for social anxiety. | Change from baseline to one-month follow-up
  Paralleling the intentions scale above, the present study developed a measure of perceived behavioral control regarding seeking treatment for social anxiety, as the existing literature lacked a sufficient and specific measure. The resulting scale includes 14 total items assessment perceived ability to seek treatment for social anxiety in the following month. Items were rated using Likert scales from 1 ("strongly disagree") to 7 ("strongly agree"), with higher scores indicating greater perceived ability to seek treatment for social anxiety.

SECONDARY OUTCOMES:
Treatment seeking behaviors | One-month follow-up
  Checklist of behavioral steps toward seeking treatment within specific domains (i.e. in-person treatment, bibliotherapy, online-treatment, medication, and alternative treatments). Because the existing literature lacks a treatment-seeking behavior questionnaire, we developed a behavioral checklist adapted from Buckner and Schmidt (2009; doi: 10.1016/j.brat.2009.04.009). The measure included 19 total treatment-seeking behaviors across the above listed domains, and as such scores could range from 0 (no steps taken toward seeking treatment since intervention) to 19 (every listed step toward every type of treatment taken since the intervention). Higher scores are considered the better outcome in the present study.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Colorado Boulder, Boulder, Colorado, United States